CLINICAL TRIAL: NCT02667626
Title: Intervening on Reproductive Health in Young Breast Cancer Survivors
Brief Title: Reproductive Health Survivorship Care Plan
Acronym: SCPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Hui-Chun Irene Su, Professor of Obstetrics, Gynecology, and Reproductive Sciences, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 140863
Record Dates: First submitted 2016-01-21; First posted 2016-01-29 (Estimated); Results first posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer; Hot Flashes; Sexual Dysfunction; Fertility; Contraception
Keywords: Breast cancer survivor; Cancer survivorship; Survivorship care plan; Vaginal dryness; Vulvovaginal atrophy; Vasomotor symptom; Infertility; Family planning
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes; Sexual Dysfunction, Physiological; Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SCPR Intervention (Experimental): Young breast cancer participants will receive their SCPR and access to additional web-based educational reproductive health information, including resource lists of helpful websites, followed by regular reproductive health prompts and study adherence reminders for 24 weeks.
  Healthcare providers of young breast cancer participants randomized to the intervention arm will receive their patient's SCPR and access to the same additional web-based educational reproductive health information as their patient, including resource lists of helpful websites.
  Interventions: Other: Reproductive Health Survivorship Care Plan (SCPR)
- Control (Active Comparator): Young breast cancer participants randomized to the waitlist control arm will receive access to the web-based resources and study adherence reminders. At completion of the 24 weeks of follow up, they will have access to their SCPR.
  Healthcare providers of young breast cancer participants randomized to the waitlist control arm will receive access to the same web-based resources as their patient.
  Interventions: Other: Control

INTERVENTIONS:
Other: Reproductive Health Survivorship Care Plan (SCPR) — The reproductive health survivorship care plan (SCPR) is a web-based educational tool that will include information on how to manage various reproductive health issues such as hot flashes, fertility concerns, contraception practices, and sexual function. The intervention also includes additional web-based information and resource lists, text-based reproductive health and study adherence prompts.
  Arms: SCPR Intervention
Other: Control — Web-based resource lists and text-based study adherence reminders
  Arms: Control

SUMMARY:
The investigators propose to test the efficacy of the Reproductive Health Survivorship Care Plan (SCP-R), a novel survivorship care tool to meet the reproductive health needs of young breast cancer survivors (YBCS). Most YBCS undergo chemotherapy and/or endocrine therapy, treatments that impair ovarian function and result in significant reproductive health late effects. These late effects include symptoms of estrogen deprivation such as hot flashes, fertility concerns, limited contraception options and sexual problems. Together they have a major, negative impact on quality of life.

Despite substantial research, treatment guidelines and clinical expertise on these issues, most YBCS and their healthcare providers have limited guidance on how best to manage these reproductive health late effects. The research team has generated a practical, accessible, evidence-based reproductive health survivorship care plan (the SCP-R) for YBCS and their providers to address this deficit in survivorship care. This clinical trial will test if YBCS who receive the web-based SCP-R are more likely than controls to improve on at least one of these reproductive health issues: hot flashes, sexual health, fertility concerns, and contraception.

DETAILED DESCRIPTION:
Participants may be recruited from throughout the United States, as all study activities may be done remotely. It is not necessary to live in San Diego or visit UC San Diego to participate in the study.

YBCS who are interested in the study will be provided access to an online screening survey to determine eligibility. Eligible YBCS who consent to the study will be followed for 24 weeks.

Following a one-week study run in, YBCS participants will be randomized to the SCPR intervention or control arms and receive the corresponding interventions.

All YBCS participants will complete 3 study time points at enrollment, 12 and 24 weeks. At each time point, they will complete a web-based study questionnaire on medical and reproductive health. YBCS participants will also daily track their hot flashes via text messaging. YBCS participants will designate a healthcare provider with whom they would discuss reproductive health issues.

Designated healthcare providers will be approached to participate in the study. Those providers who enroll will complete 2 study assessments at weeks 0 and 24. At each study time point, HCP will be assessed for preparedness on managing reproductive health issues by a web-based questionnaire.

ELIGIBILITY:
Inclusion:

* Breast cancer (Stages 0-III) diagnosis
* Breast cancer diagnosis age ≤ 45 years
* ≤ 5 years since breast cancer diagnosis
* Current age 18 to 50 years
* Completed treatment with surgery, radiation and chemotherapy (if applicable)
* Able to read English
* Able to consent to the study
* Access to an Internet connection

Exclusion:

• Women who are pregnant at recruitment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 182 (Actual)
Dates: Start 2015-03-25; Primary Completion 2017-12-31 (Actual); Study Completion 2019-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Irene Su, MD MSCE, Principal Investigator — UC San Diego
Locations (1):
- UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Interested investigators may apply for deidentified data from this study

RESULTS

PARTICIPANT FLOW:
Groups:
- SCPR Intervention: Young breast cancer participants will receive their SCPR and access to additional web-based educational reproductive health information, including resource lists of helpful websites, followed by regular reproductive health prompts and study adherence reminders for 24 weeks.
  Reproductive Health Survivorship Care Plan (SCPR): The reproductive health survivorship care plan (SCPR) is a web-based educational tool that will include information on how to manage various reproductive health issues such as hot flashes, fertility concerns, contraception practices, and sexual function. The intervention also includes additional web-based information and resource lists, text-based reproductive health and study adherence
- Control: Young breast cancer participants randomized to the waitlist control arm will receive access to the web-based resources and study adherence reminders. At completion of the 24 weeks of follow up, they will have access to their SCPR.
  Control: Web-based resource lists and text-based study adherence reminders
Period: Overall Study
Arm/Group | SCPR Intervention | Control
Started | 86 | 96
Completed | 86 | 95
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- SCPR Intervention: Young breast cancer participants will receive their SCPR and access to additional web-based educational reproductive health information, including resource lists of helpful websites, followed by regular reproductive health prompts and study adherence reminders for 24 weeks.
  Reproductive Health Survivorship Care Plan (SCPR): The reproductive health survivorship care plan (SCPR) is a web-based educational tool that will include information on how to manage various reproductive health issues such as hot flashes, fertility concerns, contraception practices, and sexual function. The intervention also includes additional web-based information and resource lists, text-based reproductive health and study adherence prompts.
- Total: Total of all reporting groups
Arm/Group | SCPR Intervention | Control | Total
Number analyzed (Participants) | 86 | 96 | 182
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 86 | 96 | 182
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (5.9) | 39.6 (6.0) | 40.0 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 96 | 182
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 82 | 90 | 172
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 7 | 8
  White | 77 | 80 | 157
  More than one race | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 86 | 96 | 182

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a 50% Decrease in Hot Flash Score
Description: 50% decrease in hot flash score. The hot flash score is calculated as the weighted sum of the number of hot flashes in each severity category multiplied by a severity-exclusive weight (1-mild, 2-moderate, 3-severe, 4-very severe). The minimum is 0 and there is no maximum. For example a woman can experience an unlimited number of hot flashes per day. Higher score indicates worse outcome.
Time Frame: Baseline and 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SCPR Intervention | Control
Number analyzed (Participants) | 86 | 96
Participants | 50 | 53

2. Primary Outcome: Number of Participants With the Reproductive Concerns After Cancer Scale - Fertility Concerns Subscale Score <=3
Description: Fertility concerns subscale score <=3. Scores for the fertility subscale calculated by averaging responses (range 1-5) to the 3 subscale questions. The minimum score is 1, the maximum score is 5, Higher scores indicate worse outcome.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SCPR Intervention | Control
Number analyzed (Participants) | 86 | 96
Participants | 24 | 14

3. Primary Outcome: Number of Participants Using a WHO Class I or II Contraception
Description: Use of World Health Organization Class I or II contraceptive methods (intrauterine devices, female sterilization, male partner sterilization, combined hormonal contraception, progestin implants or injections)
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SCPR Intervention | Control
Number analyzed (Participants) | 86 | 96
Participants | 43 | 41

4. Primary Outcome: Number of Participants With a 50% Decrease in Vulvovaginal Atrophy Score
Description: The Vulvovaginal Atrophy Score is a 4-item scale on vaginal dryness, soreness, irritation and dyspareunia experienced in the prior 4 weeks]. Each item has a 4-point Likert scale response (0-none, 1-mild, 2-moderate, 3-severe). The scale is summarized by averaging responses, with higher scores indicating a greater level of vaginal atrophy.
Time Frame: Baseline and 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SCPR Intervention | Control
Number analyzed (Participants) | 86 | 96
Participants | 37 | 39

5. Secondary Outcome: Healthcare Provider Preparedness Scale
Description: Change in score
Time Frame: 24 weeks
Population: Data were not collected
Groups:
- SCPR Intervention: Young breast cancer participants will receive their SCPR and access to additional web-based educational reproductive health information, including resource lists of websites, followed by reproductive health prompts and study adherence reminders for 24 weeks.
  Healthcare providers of young breast cancer participants randomized to the intervention arm will receive their patient's SCPR and access to the same additional web-based educational reproductive health information as their patient, including resource lists of helpful websites.
  Reproductive Health Survivorship Care Plan (SCPR): The reproductive health survivorship care plan (SCPR) is a web-based educational tool that will include information on how to manage various reproductive health issues such as hot flashes, fertility concerns, contraception practices, and sexual function. The intervention also includes additional web-based information and resource lists, text-based reproductive health and study adherence prompts.
- Control: Young breast cancer participants randomized to the waitlist control arm will receive access to the web-based resources and study adherence reminders. At completion of the 24 weeks of follow up, they will have access to their SCPR.
  Healthcare providers of young breast cancer participants randomized to the waitlist control arm will receive access to the same web-based resources as their patient.
  Control: Web-based resource lists and text-based study adherence reminders
Arm/Group | SCPR Intervention | Control
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Depression (PHQ-8)
Description: Change in score
Time Frame: 12 and 24 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Social Support (MOS Social Support)
Description: Change in score
Time Frame: 12 and 24 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Insomnia Scale
Description: Change in score
Time Frame: 12 and 24 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Female Sexual Function Inventory
Description: Change in score
Time Frame: 12 and 24 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Confidence for Managing Reproductive Health Issues Scale
Description: Change in score
Time Frame: 12 and 24 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Menopause Quality of Life (MENQOL)
Description: Change in score
Time Frame: 12 and 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | SCPR Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/96
Other Adverse Events (participants affected / at risk) | 0/86 | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT02667626/Prot_SAP_000.pdf